CLINICAL TRIAL: NCT03177564
Title: A Randomized Controlled Trial to Assess the Feasiblity of a Driving Pressure Limited Ventilation vs.Standard Strategy During Video-assisted Thoracoscopic Lobectomy
Brief Title: Driving Pressure Limited Ventilation During Video-assisted Thoracoscopic Lobectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XYFY-2017-033
Record Dates: First submitted 2017-06-04; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Complication; Thoracic Surgery
Keywords: driving pressure; one-lung ventilation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Protective Ventilation 1 (Active Comparator): Intraoperatively ventilated patients with a tidal volume (VT) of 10 ml/kg of ideal body weight, the level of PEEP at 0 cmH2O and a FiO2 of100%.
  Interventions: Procedure: Protective ventilation 1
- Protective Ventilation 2 (Active Comparator): Intraoperatively ventilated patients with a tidal volume (VT) of 6 ml/kg of ideal body weight, the level of PEEP at 5cmH2O and a FiO2 of 60% with lung recruitment maneuvers.
  Interventions: Procedure: Protective ventilation 2
- Driving Pressure Limited Ventilation (Experimental): The intervention arm receives driving pressure limited ventilation during one-lung ventilation
  Interventions: Procedure: Driving Pressure Limited Ventilation

INTERVENTIONS:
Procedure: Protective ventilation 1 — Low tidal volume, high inspired oygen fraction (FiO2) and recruitment maneuver.
  Arms: Protective Ventilation 1
Procedure: Protective ventilation 2 — Low tidal volume, PEEP, moderate inspired oygen fraction (FiO2) and recruitment maneuver.
  Arms: Protective Ventilation 2
Procedure: Driving Pressure Limited Ventilation — Positive end expiratory pressure is adjusted to minimize driving pressure, plateau pressure minus end expiratory pressure from 3 to 10 cmH2O during one-lung ventilation and a FiO2 of 60%
  Arms: Driving Pressure Limited Ventilation

SUMMARY:
This study aims to investigate the feasibility of a driving pressure limited mechanical ventilation strategy compared to a conventional strategy in patients undergoing one-lung ventilation during Video-assisted thoracoscopic lobectomy.

DETAILED DESCRIPTION:
• More recently, the so-called lung-protective intraoperative ventilation strategies have been advocated to prevent lung injury. Such strategies aim at minimizing lung hyperinflation as well as cycling collapse and reopening of lung units, through the use of low tidal volumes (VTs) and positive end-expiratory pressure (PEEP). However, despite huge improvements in surgical and anesthesia techniques and management. It is surprising that, so far, mortality and pulmonary complication rates were not reduced over time .Recently, several investigations suggest an association between high driving pressure (the difference between the plateau pressure and the level of PEEP) and outcome for patients with acute respiratory distress syndrome. It is uncertain whether a similar association exists for high driving pressure during surgery and the occurrence of postoperative pulmonary complications. In this issue, Ary S Neto and colleagues report an individual patient data meta-analysis further investigating the risk of mechanical ventilation in healthy individuals during general anesthesia .After both a multivariate and mediation analysis, the driving pressure, but not the tidal volume or the positive end-expiratory pressure applied, seemed to be the only parameter that was associated with the development of postoperative pulmonary complications. This randomized controlled trial is aims to prove that driving pressure limited ventilation is superior in preventing postoperative pulmonary complications to existing protective ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Adults greater than or equal to 18 years
2. ARISCAT（Assess Respiratory Risk in Surgical Patients in Catalonia）≥26 points
3. Patients undergoing video-assisted thoracoscopic lobectomy

Exclusion Criteria:

1. The American Society of Anesthesiologists (ASA) Physical Status classification greater than or equal to 4
2. Emergency surgery
3. Pulmonary hypertension
4. Forced vital capacity or forced expiratory volume in 1 sec < 70% of the predicted values
5. Coagulation disorder
6. Pulmonary or extrapulmonary infections
7. History of treatment with steroid in 3 months before surgery
8. History of recurrent pneumothorax
9. History of lung resection surgery
10. History of mechanical ventilation in 2 weeks
11. Body Mass Index[≥35 kg／m2 ]
12. Patient who is contraindicated with application of positive end expiratory pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-06-10 (Estimated); Study Completion 2018-06-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative pulmonary complications | within the first 3 days after surgery
  Patient is regarded to have postoperative pulmonary complication when 4 or more positive variables exists according to Melbourne Group Scale.

SECONDARY OUTCOMES:
Partial pressure of oxygen in arterial blood | 15 min after induction, 20 and 60 min after start of one-lung ventilation, 15 min after restart of two-lung ventilation, 1 hour after the end of surgery
respiratory compliance | during surgery
  Dynamic compliance, Static compliance
TNF-α | the start of one-lung ventilation, 1 hour of one-lung ventilation and the end of one-lung ventilation
IL-8 | the start of one-lung ventilation, 1 hour of one-lung ventilation and the end of one-lung ventilation
ICU mortality | Patients will be followed during the period of hospital stay, an expected average of 28 days
In-hospital mortality | Patients will be followed during the period of hospital stay, an expected average of 28 days
28-day survival | From day 0 to day 28

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neto AS, Hemmes SN, Barbas CS, Beiderlinden M, Fernandez-Bustamante A, Futier E, Gajic O, El-Tahan MR, Ghamdi AA, Gunay E, Jaber S, Kokulu S, Kozian A, Licker M, Lin WQ, Maslow AD, Memtsoudis SG, Reis Miranda D, Moine P, Ng T, Paparella D, Ranieri VM, Scavonetto F, Schilling T, Selmo G, Severgnini P, Sprung J, Sundar S, Talmor D, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Amato MB, Costa EL, de Abreu MG, Pelosi P, Schultz MJ; PROVE Network Investigators. Association between driving pressure and development of postoperative pulmonary complications in patients undergoing mechanical ventilation for general anaesthesia: a meta-analysis of individual patient data. Lancet Respir Med. 2016 Apr;4(4):272-80. doi: 10.1016/S2213-2600(16)00057-6. Epub 2016 Mar 4. PMID 26947624
- [Result] Mazo V, Sabate S, Canet J, Gallart L, de Abreu MG, Belda J, Langeron O, Hoeft A, Pelosi P. Prospective external validation of a predictive score for postoperative pulmonary complications. Anesthesiology. 2014 Aug;121(2):219-31. doi: 10.1097/ALN.0000000000000334. PMID 24901240
- [Result] Agostini P, Cieslik H, Rathinam S, Bishay E, Kalkat MS, Rajesh PB, Steyn RS, Singh S, Naidu B. Postoperative pulmonary complications following thoracic surgery: are there any modifiable risk factors? Thorax. 2010 Sep;65(9):815-8. doi: 10.1136/thx.2009.123083. PMID 20805178
- [Result] Hager DN. Recent Advances in the Management of the Acute Respiratory Distress Syndrome. Clin Chest Med. 2015 Sep;36(3):481-96. doi: 10.1016/j.ccm.2015.05.002. Epub 2015 Jul 2. PMID 26304285
- [Result] Guerin C, Papazian L, Reignier J, Ayzac L, Loundou A, Forel JM; investigators of the Acurasys and Proseva trials. Effect of driving pressure on mortality in ARDS patients during lung protective mechanical ventilation in two randomized controlled trials. Crit Care. 2016 Nov 29;20(1):384. doi: 10.1186/s13054-016-1556-2. PMID 27894328
- [Result] Loring SH, Malhotra A. Driving pressure and respiratory mechanics in ARDS. N Engl J Med. 2015 Feb 19;372(8):776-7. doi: 10.1056/NEJMe1414218. No abstract available. PMID 25693019
- [Result] Xie J, Jin F, Pan C, Liu S, Liu L, Xu J, Yang Y, Qiu H. The effects of low tidal ventilation on lung strain correlate with respiratory system compliance. Crit Care. 2017 Feb 3;21(1):23. doi: 10.1186/s13054-017-1600-x. PMID 28159013
- [Result] Grieco DL, Chen L, Dres M, Brochard L. Should we use driving pressure to set tidal volume? Curr Opin Crit Care. 2017 Feb;23(1):38-44. doi: 10.1097/MCC.0000000000000377. PMID 27875410